CLINICAL TRIAL: NCT01262716
Title: A Novel Therapy for the Treatment of Chest Wall Progression of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Rogers Sciences Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Tufts Medical Center (Other)
Responsible Party: Samuel L Hill, Rogers Sciences Inc.
Other Study IDs: 9439; R43CA139644-01A1 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: Chest wall progression breast cancer; PDT; Photofrin; Photosensitizer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will assess safety and ergonomics/engineering design of a novel cancer treatment, Continuous Low Irradiance Photodynamic therapy (CLIPT). We will assess the effects on primary and metastatic tumors involving the skin, in particular to improve the functionality, efficiency and wearability of the light delivery device (LDD) as well as the overall treatment in subjects with chest wall recurrences of breast cancer. An ongoing study (IRB# 8227), sponsored by a Susan G. Komen Breast Cancer Foundation grant, using a 1st generation LDD device has evaluated and determined a dose-limiting toxicity of CLIPT for subjects with chest wall recurrences of breast cancer.

A Diomed laser will be the device used in this study. The Diomed laser will deliver 630 nm (red spectrum) light through a Fiber Optic Patch. The Fiber Optic patch will be compatible with the laser, delivering light to a designated region on the patient's skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age, with primary or metastatic cutaneous tumors that may or may not have been previously irradiated.
* ECOG performance status < 3.
* Patients must not have received any systemic anti-cancer therapy within 30 days prior to enrolling in this study.
* Patients must not have received radiation therapy to the target site within 60 days of enrolling on this study.
* Skin of target site and control site must be grade 0 or 1 by Common Terminology
* Patients must have a target lesion and normal peri-umbilical skin that can be covered by the fiber-optic mesh used to deliver CLIPT (10 x 10 cm, or 3 x 3).
* If located on an extremity, the target lesion must not cover more than 50% of the diameter of the extremity at the level at which it is located.
* Absolute neutrophil count > 1000.
* Adequate coagulation status as indicated by platelet count > 50,000, PT and PTT < 1.5 time the upper limit of normal.
* Patients must sign informed consent.

Exclusion Criteria:

* Male patients not considered for this study.
* Patients must have a target lesion in a location other than the hands, feet, genitals, or face. Lesions in those locations will be excluded.
* Patients with medical conditions associated with photosensitivity, such as cutaneous porphyria or a collagen vascular disease, or with known allergies to porphyrins will be excluded.
* Pregnant and nursing patients will be excluded. Women of child-bearing potential must have a negative serum or urine pregnancy test prior to enrollment.
* Patients taking medications known to cause photosensitivity (tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics, griseofulvin, and fluoroquinolones, St. John's wort and amiodarone) will be excluded.
* Patients with severe hepatic dysfunction (total bilirubin, AST, or ALT > five times upper limit of normal) will be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of 3 female patients. Eligible patients will be recruited from cancer centers in North America specializing in breast cancer. Recruitment has begun with the Hematology/Oncology, Dermatologic Oncology, and Radiation Oncology programs at Tufts Medical Center, Rhode Island Hospital and the teaching hospitals affiliated with Tufts and Brown Universities. All research related activity will only take place at the Tufts Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary S. Rogers, M.D., Study Director — Rogers Sciences Inc.; Roger A. Graham, M.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States